CLINICAL TRIAL: NCT00170612
Title: A Single-Blind Open-Label Randomized Phase II Study of the Safety, Immunogenicity and Impact on Pneumococcus (Pnc) Carriage of the Pnc Vaccination Regimens Combining 1, 2, or 3 Doses of 7-Valent Pneumococcal Conjugate Vaccine (PCV) in the First 4 Months of Life Followed by a Single Dose of 23-Valent Pneumococcal Polysaccharide Vaccine (PPS) at 12 Months of Age
Brief Title: Pneumococcal Vaccination of Fiji Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Fiona Russell, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 03-042; FNRERC Reference # 2002-001
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Pneumococcal Infections
Keywords: Pneumococcal infections; Fiji; infants; vaccine
MeSH Terms: conditions — Pneumococcal Infections | interventions — 23-valent pneumococcal capsular polysaccharide vaccine; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- A (Experimental): PCV at 6 weeks, 10 weeks, and 14 weeks; PPS at 18 months
  Interventions: Biological: Pneumovax 23; Biological: Prevnar
- B (Experimental): PCV at 6 weeks, 10 weeks, and 14 weeks; PPS at 12 months and 18 months
  Interventions: Biological: Pneumovax 23; Biological: Prevnar
- C (Experimental): PCV at 6 weeks and 14 weeks; PPS at 18 months
  Interventions: Biological: Pneumovax 23; Biological: Prevnar
- D (Experimental): PCV at 6 weeks and 14 weeks; PPS at 12 months and 18 months
  Interventions: Biological: Pneumovax 23; Biological: Prevnar
- E (Experimental): PCV at 14 weeks; PPS at 18 months
  Interventions: Biological: Pneumovax 23; Biological: Prevnar
- F (Experimental): PCV at 14 weeks; PPS at 12 months and 18 months
  Interventions: Biological: Pneumovax 23; Biological: Prevnar
- G (Experimental): No PCV; PPS at 12 months and 18 months
  Interventions: Biological: Pneumovax 23
- H (Active Comparator): No PCV; PPS at 18 months
  Interventions: Biological: Pneumovax 23

INTERVENTIONS:
Biological: Pneumovax 23 — 23-valent PPS, 25 micrograms/serotype
Biological: Prevnar — 7-valent PCV, 2 micrograms/serotype, except serotype 6B which is 4 micrograms/serotype
  Arms: A; B; C; D; E; F

SUMMARY:
Pneumonia is the most common reason for admission of Fijian children to hospitals. The most common germ causing pneumonia is "streptococcus pneumoniae." It is a common cause of meningitis (infection around the brain and spinal cord), ear infections, and blood infections and it lives in the nose of humans. A vaccine has been developed that will help prevent these common diseases but prevents only about one quarter of pneumonia cases and it is expensive. This study explores new ways of giving this vaccine that are affordable, safe, and effective in countries such as Fiji. About 550 Fijian infants presenting at 6 weeks of age, for their first diptheria, tetanus, toxoid, pertussis vaccine immunization, to one of the participating Health Centers or Colonial War Memorial Hospital in urban Suva, Fiji will be enrolled. Children will remain in the study for 2 years. Study procedures include full vaccination against 7 types of pneumococcus, blood tests, and nasal swabs.

DETAILED DESCRIPTION:
This research project began as a study of alternative strategies for Pnc (Pneumococcus) immunization for children in developing countries. In the original study, infants presenting to a health center in urban Fiji were randomized to receive 1, 2, or 3 doses of PCV (Prevnar) followed by a dose of 23-valent PPS (Pneumococcal polysaccharide vaccine) at 6 or 9 months of age. The regimens were compared with each other and with 2 control groups with respect to immunogenicity, impact on carriage of vaccine type Pnc, and response to a small dose of PPS at 15 months of age. After the trial was underway and 228 infants had been recruited, concerns were raised about the safety of PPS in infancy. Specifically concerns were raised that it might result in later immunological hyporesponsiveness in some of the recipients, to some of the serotypes. After a thorough review it was decided to proceed with the study, but to modify it so that it addressed directly the issue of potential hyporesponsiveness, while not giving PPS to any children under 12 months of age. This protocol represents the completion of the study with the new design for the children already enrolled, and a new design for a further cohort of children who will be enrolled. The newly designed trial will be a single blind, open-label, randomized, controlled trial of 550 healthy infants. Infants will be randomized to 1 of 8 equal groups to receive 0, 1, 2, or 3 doses of PCV (Pneumococcal conjugate vaccine), with or without a booster of PPS at 12 months of age. Two control groups will be recruited, 1 will receive no PCV in infancy and the other will receive a dose of PPS at 12 months of age. At 18 months of age, all infants will receive a 20 percent dose of PPS to stimulate and allow the assessment of immunological memory. At 2 years of age, any child who has received no or one dose of PCV (Groups E, F, G and H) will receive a single dose of PCV. Blood samples will be taken at 18 weeks age, 12 months of age, before the 18 months dose and 4 weeks later. In addition half of the children will have a blood sample taken at 9 months and the other half will have a sample taken 2 weeks after their 12 month dose of PPS. The 9- and 12-month blood sample will assess the long-term persistence of circulating antibody and avidity maturation following a 1, 2, or 3 dose primary series of PCV. The primary objective is to demonstrate noninferiority at 19 months of age, of those groups receiving PPS at 12 months and those who do not with respect to the proportion of children in each group, with a satisfactory immune response at 19 months of age, measured by OPA to each of the 11 serotypes included in the PPS for which an OPA has been developed. The secondary objective is to assess the immunogenicity and impact on carriage of various Pnc vaccination regimens that combine 1 to 3 doses of PCV with a dose of PPS, concerns regarding the potential for the development of hyporesponsiveness. Endpoints to be evaluated will include serotype specific immunoglobulin G antibody measured by enzyme-linked immunosorbent assay to the 23 serotypes in the PPS, avidity assays to the same serotypes, opsonophagocytic assays to the 11 serotypes for which these assays are currently available, and Pnc carriage by serotype. With hyporesponsiveness as the primary endpoint of interest a scheme of analysis has been proposed which will require a minimum sample size of 500.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infant aged between 6 and 8 weeks
2. No significant maternal or perinatal history
3. Written and signed parental/caregiver consent
4. Lives within 30 minutes of the health clinic
5. Family anticipate living in the study area for the next 2 years

Exclusion Criteria:

1. Known allergy to any component of the vaccine
2. Allergic reaction or anaphylactoid reaction with previous vaccines
3. Known immunodeficiency disorder
4. HIV positive mother (many women are tested for HIV antenatally, however a test is not planned; therefore it would be based on clinic records or self report)
5. Known thrombocytopenia or coagulation disorder
6. On immunosuppressive medication
7. Received any blood product since birth
8. Severe congenital anomaly
9. Chronic or progressive disease
10. Seizure disorder
11. History of invasive Pneumococcal, meningococcal, or Haemophilus influenzae diseases
12. Moderate or severe acute infection (temporary exclusion); Minor illnesses such as an uncomplicated upper respiratory tract infection, localized skin infections, or mild diarrhea will not be an exclusion criterion

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 552 (Actual)
Dates: Start 2005-11; Primary Completion 2008-01 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
For each serotype assayed (23 for ELISA and 11 for functional assays) the proportion of children responding to the micro-PPS dose at 18 months and the GMC of the response will be compared between children who receive PPS at 12 months and those who do not | 19 months of age

SECONDARY OUTCOMES:
Proportion of children showing hyporesponse at 18 months to more than half of all 23 serotypes | 18 weeks; 12.5 months of age
Immunogenicity and carriage: Immune responses following the primary series of conjugate vaccination, measured by ELISA and OPA will be compared between the group receiving two doses of PCV and those receiving 3 doses of vaccine | 18 months of age
Rate of decline: assessment of antibody levels | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Fiona M Russell, FRACP, Principal Investigator — University of Melbourne
Locations (1):
- Colonial War Memorial Hospital, Suva, Fiji

REFERENCES:
- [Derived] Russell FM, Balloch A, Licciardi PV, Carapetis JR, Tikoduadua L, Waqatakirewa L, Cheung YB, Mulholland EK, Tang ML. Serotype-specific avidity is achieved following a single dose of the 7-valent pneumococcal conjugate vaccine, and is enhanced by 23-valent pneumococcal polysaccharide booster at 12 months. Vaccine. 2011 Jun 15;29(27):4499-506. doi: 10.1016/j.vaccine.2011.04.038. Epub 2011 May 1. PMID 21539882
- [Derived] Russell FM, Carapetis JR, Burton RL, Lin J, Licciardi PV, Balloch A, Tikoduadua L, Waqatakirewa L, Cheung YB, Tang ML, Nahm MH, Mulholland EK. Opsonophagocytic activity following a reduced dose 7-valent pneumococcal conjugate vaccine infant primary series and 23-valent pneumococcal polysaccharide vaccine at 12 months of age. Vaccine. 2011 Jan 10;29(3):535-44. doi: 10.1016/j.vaccine.2010.10.046. Epub 2010 Oct 31. PMID 21044669
- [Derived] Russell FM, Carapetis JR, Satzke C, Tikoduadua L, Waqatakirewa L, Chandra R, Seduadua A, Oftadeh S, Cheung YB, Gilbert GL, Mulholland EK. Pneumococcal nasopharyngeal carriage following reduced doses of a 7-valent pneumococcal conjugate vaccine and a 23-valent pneumococcal polysaccharide vaccine booster. Clin Vaccine Immunol. 2010 Dec;17(12):1970-6. doi: 10.1128/CVI.00117-10. Epub 2010 Oct 13. PMID 20943882
- [Derived] Russell FM, Carapetis JR, Balloch A, Licciardi PV, Jenney AW, Tikoduadua L, Waqatakirewa L, Pryor J, Nelson J, Byrnes GB, Cheung YB, Tang ML, Mulholland EK. Hyporesponsiveness to re-challenge dose following pneumococcal polysaccharide vaccine at 12 months of age, a randomized controlled trial. Vaccine. 2010 Apr 26;28(19):3341-9. doi: 10.1016/j.vaccine.2010.02.087. Epub 2010 Mar 4. PMID 20206670
- [Derived] Russell FM, Licciardi PV, Balloch A, Biaukula V, Tikoduadua L, Carapetis JR, Nelson J, Jenney AW, Waqatakirewa L, Colquhoun S, Cheung YB, Tang ML, Mulholland EK. Safety and immunogenicity of the 23-valent pneumococcal polysaccharide vaccine at 12 months of age, following one, two, or three doses of the 7-valent pneumococcal conjugate vaccine in infancy. Vaccine. 2010 Apr 19;28(18):3086-94. doi: 10.1016/j.vaccine.2010.02.065. Epub 2010 Mar 1. PMID 20199764